CLINICAL TRIAL: NCT01703988
Title: An Open-Label, Dose Escalation Study to Assess the Safety, Tolerability and Dose-Range Finding of Multiple Doses of ISIS 396443 Delivered Intrathecally to Patients With Spinal Muscular Atrophy
Brief Title: An Open-label Safety, Tolerability and Dose-Range Finding Study of Multiple Doses of Nusinersen (ISIS 396443) in Participants With Spinal Muscular Atrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 396443 - CS2; 2017-000327-27 (EudraCT Number)
Expanded Access: NCT02865109 (No longer available)
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; SMA; SMN; SMNRx; ISIS-SMNRx; ISIS 396443
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nusinersen 3 mg (Experimental): 3 mg nusinersen on Days 1, 29, 85, intrathecal (IT) injection
  Interventions: Drug: Nusinersen
- Nusinersen 6 mg (Experimental): 6 mg nusinersen on Days 1, 29, 85, IT injection
  Interventions: Drug: Nusinersen
- Nusinersen 9 mg (Experimental): 9 mg nusinersen on Days 1 and 85, IT injection
  Interventions: Drug: Nusinersen
- Nusinersen 12 mg (Experimental): 12 mg nusinersen on Days 1, 29, 85, IT injection
  Interventions: Drug: Nusinersen

INTERVENTIONS:
Drug: Nusinersen — Single IT injection for each dose
  Other Names: ISIS-SMNRx; ISIS 396443; BIIB058; Spinraza

SUMMARY:
This study will test the safety, tolerability, and pharmacokinetics of escalating doses of nusinersen (ISIS 396443) administered into the spinal fluid either two or three times over the duration of the trial, in participants with spinal muscular atrophy (SMA).

Four dose levels will be evaluated sequentially. Each dose level will be studied in a cohort of approximately 8 participants, where all participants will receive active drug.

DETAILED DESCRIPTION:
This study was conducted and the protocol was registered by Ionis Pharmaceuticals, Inc. In August 2016, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Genetic documentation of 5q SMA (homozygous gene deletion or mutation)
* Clinical signs attributable to SMA
* Able to complete all study procedures, measurements, and visits and parent/patient has adequately supportive psychosocial circumstances, in the opinion of the Investigator
* Estimated life expectancy > 2 years from Screening
* Meets age-appropriate institutional criteria for use of anesthesia/sedation, if use is planned for study procedure

Key Exclusion Criteria:

* Respiratory insufficiency defined by the medical necessity for invasive or non-invasive ventilation during a 24-hour period
* Medical necessity for a gastric feeding tube, where the majority of feeds are given by this route, as assessed by the Investigator
* Previous scoliosis surgery that would interfere with the lumbar puncture injection procedure
* Hospitalization for surgery (e.g. scoliosis surgery) or pulmonary event within 2 months of screening or planned during the duration of the study
* Presence of an untreated or inadequately treated active infection requiring systemic antiviral or antimicrobial therapy at any time during the screening period
* History of brain or spinal cord disease that would interfere with lumbar puncture procedures or cerebrospinal fluid (CSF) circulation
* Presence of an implanted shunt for the drainage of CSF or an implanted central nervous system catheter
* History of bacterial meningitis
* Dosing with ISIS 396443 in clinical study ISIS 396443-CS1 Cohorts 2, 3, or 4
* Dosing with ISIS 396443 in clinical study ISIS 396443-CS10
* Clinically significant abnormalities in hematology or clinical chemistry parameters or electrocardiogram (ECG) at the Screening visit, as assessed by the Site Investigator that would render the subject unsuitable for inclusion
* Treatment with investigational drug, biological agent, or device within 1-month of Screening or 5 half-lives of study agent, whichever is longer. Treatment with valproate or hydroxyurea within 3-months of screening. Any history of gene therapy or cell transplantation
* Ongoing medical condition that would interfere with the conduct and assessments of the study. Examples are medical disability (e.g. wasting or cachexia, severe anemia) that would interfere with the assessment of safety or would compromise the ability of the patient to undergo study procedures.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2012-10-31 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (4):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - UT Southwestern Medical Center - Children's Medical Center Dallas, Dallas, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Darras BT, Farrar MA, Mercuri E, Finkel RS, Foster R, Hughes SG, Bhan I, Farwell W, Gheuens S. An Integrated Safety Analysis of Infants and Children with Symptomatic Spinal Muscular Atrophy (SMA) Treated with Nusinersen in Seven Clinical Trials. CNS Drugs. 2019 Sep;33(9):919-932. doi: 10.1007/s40263-019-00656-w. PMID 31420846
- See also: Clinical Study Report (CSR) Synopsis - a results summary — http://clinicalresearch.biogen.com/Content/Studies/CS2%20Biogen.com%20Packet.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nusinersen 3 mg | Nusinersen 6 mg | Nusinersen 9 mg | Nusinersen 12 mg
Started | 8 | 8 | 9 | 9
Completed | 8 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 1
Not completed — Investigator Judgment | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Nusinersen 3 mg: 3 mg nusinersen on Days 1, 29, 85, IT injection
- Total: Total of all reporting groups
Arm/Group | Nusinersen 3 mg | Nusinersen 6 mg | Nusinersen 9 mg | Nusinersen 12 mg | Total
Number analyzed (Participants) | 8 | 8 | 9 | 9 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (5.4) | 8.1 (5.2) | 6.0 (4.0) | 6.9 (4.3) | 7.4 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 3 | 14
  Male | 4 | 5 | 5 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Discontinuations Due to AEs, and Highest Severity of AEs
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the study or use of the investigational drug product, whether or not the AE is considered related to the investigational drug product. An SAE is any AE that, in the view of either the Investigator or Sponsor, meets any of the following criteria: results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly or birth defect; and is an important medical event in the judgment of the investigator. Drug-related is an event related or possibly related to study drug. Severity of AEs was assessed as mild, moderate, or severe.
Time Frame: Participants were followed for the duration of the study; mean (SD) duration of treatment was 82.9 (15.4) days
Population: Safety Population, defined as all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Nusinersen 3 mg | Nusinersen 6 mg | Nusinersen 9 mg | Nusinersen 12 mg
Number analyzed (Participants) | 8 | 8 | 9 | 9
Participants
  Any AE | 8 | 6 | 9 | 9
  Any drug-related AE | 0 | 0 | 0 | 0
  Any SAE | 2 | 0 | 0 | 1
  Discontinued due to an AE | 0 | 0 | 0 | 0
  Highest severity of AE=mild | 2 | 2 | 6 | 5
  Highest severity of AE=moderate | 4 | 2 | 3 | 4
  Highest severity of AE=severe | 2 | 2 | 0 | 0

2. Secondary Outcome: Plasma Pharmacokinetics: Maximal Observed Plasma Drug Concentration (Cmax)
Time Frame: Day 1 and Day 85
Population: Pharmacokinetic (PK) Population, defined as all enrolled participants who have evaluable PK data; number analyzed=participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nusinersen 3 mg | Nusinersen 6 mg | Nusinersen 9 mg | Nusinersen 12 mg
Number analyzed (Participants) | 8 | 8 | 9 | 9
ng/mL
  Day 1 | 51.5 (72.7) | 79.8 (57.2) | 141.0 (52.8) | 208.0 (110.0)
  Day 85: number analyzed (Participants) | 8 | 8 | 9 | 8
  Day 85 | 32.5 (32.3) | 52.8 (33.5) | 127.0 (37.7) | 132.0 (85.6)

3. Secondary Outcome: Plasma Pharmacokinetics: Time to Reach Cmax in Plasma
Time Frame: Day 1 and Day 85
Population: PK Population, defined as all enrolled participants who have evaluable PK data; number analyzed=participants with an assessment at given time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Nusinersen 3 mg | Nusinersen 6 mg | Nusinersen 9 mg | Nusinersen 12 mg
Number analyzed (Participants) | 8 | 8 | 9 | 9
hours
  Day 1 | 5.09 [2.03 to 12.0] | 5.93 [2.00 to 23.0] | 3.92 [2.00 to 8.03] | 4.05 [1.97 to 12.0]
  Day 85: number analyzed (Participants) | 8 | 8 | 9 | 8
  Day 85 | 6.08 [4.12 to 6.17] | 6.04 [5.97 to 6.25] | 4.12 [2.00 to 6.25] | 5.92 [1.95 to 6.07]

4. Secondary Outcome: Plasma Pharmacokinetics: Plasma Pharmacokinetics: Area Under the Plasma Concentration Time Curve From the Time of the IT Dose to 6 Hours After Dosing (AUC0-6hr)
Time Frame: Day 1 and Day 85
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Nusinersen 3 mg | Nusinersen 6 mg | Nusinersen 9 mg | Nusinersen 12 mg
Number analyzed (Participants) | 8 | 8 | 9 | 9
ng*hr/mL
  Day 1 | 181 (225) | 306 (259) | 601 (249) | 823 (442)
  Day 85: number analyzed (Participants) | 8 | 8 | 9 | 8
  Day 85 | 110 (107) | 179 (135) | 524 (185) | 555 (398)

5. Secondary Outcome: Cerebrospinal Fluid (CSF) Pharmacokinetics: Predose CSF Drug Concentrations
Time Frame: Day 1, Day 29, and Day 85
Population: PK Population, defined as all enrolled participants who have evaluable PK data; number analyzed=participants with an assessment at given time point. (This study includes participants previously enrolled in Study ISIS 396443 - CS1 (NCT01494701).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nusinersen 3 mg | Nusinersen 6 mg | Nusinersen 9 mg | Nusinersen 12 mg
Number analyzed (Participants) | 8 | 8 | 9 | 9
ng/mL
  Day 1: number analyzed (Participants) | 6 | 8 | 6 | 9
  Day 1 | 0.0651 (0.117) | 0.0560 (0.104) | NA (NA) — below the limit of quantification (50 pg/mL) | NA (NA) — below the limit of quantification (50 pg/mL)
  Day 29: number analyzed (Participants) | 7 | 8 | 0 | 7
  Day 29 | 1.41 (0.456) | 2.65 (1.44) |  | 2.22 (0.924)
  Day 85: number analyzed (Participants) | 8 | 8 | 9 | 7
  Day 85 | 2.12 (0.573) | 3.76 (2.05) | 1.50 (0.447) | 3.36 (1.04)

6. Secondary Outcome: Urine Pharmacokinetics: Renal Clearance, Cohort 4
Description: Renal clearance of nusinersen for participants was assessed in the 12 mg reporting group only, per protocol.
Time Frame: Day 1 and Day 85
Population: Pharmacokinetic (PK) Population, defined as all enrolled participants who have evaluable PK data
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Nusinersen 12 mg
Number analyzed (Participants) | 6
mL/hr
  Day 1 | 0.674 (0.602)
  Day 85 | 77.5 (92.5)

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of the study; mean (SD) duration of treatment was 82.9 (15.4) days.
Description: Treatment emergent AEs are presented regardless of seriousness or relationship to investigational product.
Arm/Group | Nusinersen 3 mg | Nusinersen 6 mg | Nusinersen 9 mg | Nusinersen 12 mg
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/8 | 0/9 | 1/9
Other Adverse Events (participants affected / at risk) | 8/8 | 6/8 | 9/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nusinersen 3 mg (N=8) | Nusinersen 6 mg (N=8) | Nusinersen 9 mg (N=9) | Nusinersen 12 mg (N=9)
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 — Event assessed as unlikely to be related to study drug.
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nusinersen 3 mg (N=8) | Nusinersen 6 mg (N=8) | Nusinersen 9 mg (N=9) | Nusinersen 12 mg (N=9)
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1
Strabismus (Eye disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Puncture site pain (General disorders) | 0 | 3 | 3 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 3
Fatigue (General disorders) | 1 | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 1
Catheter site related reaction (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0
Gravitational oedema (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2 | 1
Pharyngitis streptococcal (Infections and infestations) | 3 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 0
Localised infection (Infections and infestations) | 0 | 0 | 2 | 0
Otitis media (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Eye infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 3 | 1 | 3 | 5
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Torus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Agitation postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 4
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pelvic deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 2 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Dyslexia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysphoria (Psychiatric disorders) | 1 | 0 | 0 | 0
Parasomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.